CLINICAL TRIAL: NCT00814814
Title: Protein S100 Beta as a Predictor of the Outcome of Cardiopulmonary Resuscitation
Brief Title: Protein S100 Beta as a Predictor of Resuscitation Outcome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr Sharon Einav, Dr., Shaare Zedek Medical Center
Other Study IDs: 14-01-05 A and B (correction)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Cardiopulmonary Arrest Outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiopulmonary arrest

SUMMARY:
Management of cardiac arrest is complicated by the lack of a readily available tool identifying individuals who are likely to be successfully resuscitated. S100 beta is a protein that originates in the astroglial cells of the brain, and NSE (Neuron Specific Enolase) is another protein that originates in the neurons themselves. In the laboratory, the concentration of these proteins correlate with evidence of brain damage after head trauma, stroke and exposure to low levels of oxygen. The concentration of these proteins in the blood of human survivors of cardiopulmonary resuscitation in humans is much higher than in patients who were resuscitated but did not survive. However, it is still unclear whether survivors from cardiopulmonary resuscitation have higher levels of these proteins in their blood if they survive with neurological injury secondary to the arrest and resuscitation.

Hypothesis: In humans, the blood concentrations of protein S100 beta and NSE during and after resuscitation can predict who will die despite cardiopulmonary resuscitation and who will survive with neurological injury secondary to the arrest and resuscitation.

ELIGIBILITY:
Inclusion Criteria:

* All victims of non-traumatic out-of hospital cardiopulmonary arrest (defined as the absence of either spontaneous respiration or palpable pulse or both) within the Jerusalem district.

Exclusion Criteria:

* Patients with do-not-resuscitate orders or an advance directive to that effect.
* Patients with intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All victims of non-traumatic out-of hospital cardiopulmonary arrest (defined as the absence of either spontaneous respiration or palpable pulse or both) within the Jerusalem district.
Sampling Method: Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2008-02; Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Poor versus good patient outcome at discharge was used to test the study hypotheses of improved prediction attributable to S100B and NSE concentration. | within 24 hours of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Einav, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (2):
- Israel (2):
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Einav S, Kaufman N, Algur N, Strauss-Liviatan N, Kark JD. Brain biomarkers and management of uncertainty in predicting outcome of cardiopulmonary resuscitation: a nomogram paints a thousand words. Resuscitation. 2013 Aug;84(8):1083-8. doi: 10.1016/j.resuscitation.2013.01.031. Epub 2013 Feb 4. PMID 23391666
- [Result] Einav S, Kaufman N, Algur N, Kark JD. Modeling serum biomarkers S100 beta and neuron-specific enolase as predictors of outcome after out-of-hospital cardiac arrest: an aid to clinical decision making. J Am Coll Cardiol. 2012 Jul 24;60(4):304-11. doi: 10.1016/j.jacc.2012.04.020. PMID 22813607